CLINICAL TRIAL: NCT04118192
Title: Can Patients With Residual Cancer After Chemotherapy for Early Breast Cancer be Identified With Multiple Ultrasound-guided Biopsies?
Brief Title: NOSTRA-Feasibility Study: A Study Looking at Ultrasound Guided Biopsies for Breast Cancer
Acronym: NOSTRA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Roche Pharma AG (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: RG_16-108
Record Dates: First submitted 2019-09-05; First posted 2019-10-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; HER2 positive; ER negative; Tumour bed core biopsies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour bed core biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tumour bed core biopsy — Collection of up to 8 core biopsies across 4 zones of the whole tumour bed to detect residual cancer post neo-adjuvant treatment

SUMMARY:
A prospective non-randomised multi-centre feasibility study to assess if patients with residual cancer following dual-targeted neoadjuvant chemotherapy treatment for HER2-positive, ER-negative early breast cancer can be identified by multiple ultrasound (US)-guided tumour bed core biopsies

DETAILED DESCRIPTION:
The NOSTRA-Feasibility study is designed to determine if it is safe to omit surgery after the planned neoadjuvant chemotherapy plus dual-targeted anti-HER2 treatment. The study is needed to determine whether patients with residual cancer can be identified by histological examination of multiple ultrasound-guided tumour bed core biopsies following dual-targeted neoadjuvant treatment for HER2-positive, ER-negative early primary breast cancer and whether there is concordance between local pathology reporting and central pathology reporting by the trials expert pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histological diagnosis of operable HER2-positive, ER-negative, early stage invasive breast cancer
* Tumour size ≥ 1cm and visible on US (T1c to T4d)
* Patient fit and willing to receive, or is already receiving and has received no more than five cycles of a NOSTRA-Feasibility Study approved treatment regimen, in the opinion of the responsible clinician
* Eastern Co-operative Group (ECOG) performance status of 0 or 1
* Women of child-bearing potential, prepared to adopt highly effective contraceptive measures if sexually active for at least 6 months after completion of study medication
* Female, 18 years or older
* Able to provide informed consent for the study
* Availability of embedded paraffin tumour blocks from pre-chemotherapy biopsy
* The radiology team are able and willing to perform the tumour bed core biopsies

Exclusion Criteria:

* Previous ipsilateral invasive breast cancer or Ductal Carcinoma in Situ (DCIS)
* Unequivocal evidence of distant metastatic disease at registration
* Multi-focal disease at diagnosis
* Active malignancy
* Previous chemotherapy
* Prior extensive radiotherapy (as judged by the Investigator) to bone marrow
* Risk factors precluding the safe administration of the intended cytotoxic chemotherapy regimen
* Patient unsuitable for the planned dual-targeted anti-HER2 treatment in opinion of the Investigator
* Prior diagnosis of cardiac failure
* Uncontrolled hypertension, coronary heart disease or other significant cardiac abnormality
* Bleeding diathesis
* Any evidence of other disease which in the opinion of the Investigator places the patient at high risk of treatment related complications
* Pregnant (female patients of child bearing potential must have a urine or blood Human Chorionic Gonadotropin test performed to rule out pregnancy prior to study entry)
* Patient lactating
* Patients who have received live vaccine within 4 weeks of the date of study entry
* Any concomitant medical or psychiatric problems which in the opinion of the Investigator would prevent completion of treatment or follow-up
* Patient unfit and/or unwilling to undergo surgery
* Patient unwilling or unable to comply with scheduled visits, treatment plan and study procedures
* Patient has started protocol non-compliant neo-adjuvant chemotherapy
* Patient has started approved neoadjuvant chemotherapy but insufficient data is available to complete relevant CRFs
* Patient has already received more than five cycles of approved neoadjuvant chemotherapy

Additional Inclusion Criteria for ctDNA Sub-Study

* Patient has not yet started neoadjuvant treatment
* Patient is willing and able to give blood samples as per ctDNA Sub-Study Guidelines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER-2 positive ER-negative breast cancer patients
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Observed number of patients with false negative biopsies | 12 months post last patient recruited
  The observed number of patients with false negative biopsies (i.e. no tumour in the biopsy but tumour in the surgical specimen) as a proportion of all those assessed by Local Histopathology Review.

SECONDARY OUTCOMES:
Concordance between Local and Central Histopathology Review of core biopsies | 12 months post last patient recruited
  The number of patients whose initial local pathological assessment of pCR is confirmed by Central Histopathology Review.
Compliance with treatment | 12 months post last patient recruited
  Assessed by calculating relative dose intensity taking into account both reductions in dose and delays to treatment.
Time to local recurrence | Number of days from registration to local recurrence (if within trial duration, approximately 1.5 years)
  Defined in whole days from date of registration to local recurrence or death from any cause. Patients who are alive and without local recurrence at the time of analysis will be censored at the date last seen.
Time to distant recurrence | Number of days from registration to distant recurrence (if within trial duration, approximately 1.5 years)
  Defined in whole days from date of registration to distant recurrence or death from any cause. Patients who are alive and without distant recurrence at the time of analysis will be censored at the date last known to be alive.
Overall survival | Whole days from registration to death from any cause (if within trial duration, approximately 1.5 years)
  Defined in whole days as the date of registration to death from any cause. Patients alive at the time of analysis will be censored at the date last seen.
Re-evaluation of the primary outcome using the Central Pathological Review determination of RCB to define false negative biopsies as RCB-0 or 1 (i.e. no tumour or minimal residual disease) in the core biopsies but RCB-2 or 3 in the surgical specimen | Post-last patient last surgery (within approximately 1.5 years of start of trial)
  This will be reported as a proportion of all recruited patients.
Ability of the axillary lymph node assessments post-neoadjuvant treatment to identify definitive axillary lymph node involvement determined by surgery histopathology | Post-last patient last surgery (within approximately 1.5 years of start of trial)
  Sensitivity, specificity and false negative rates will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rea, Principal Investigator — University of Birmingham
Locations (24):
- United Kingdom (24):
  - Basildon Hospital, Basildon, Essex
  - Belfast City Hospital, Belfast
  - City Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Blackpool Teaching Hospitals NHS Trust, Blackpool
  - Southmead Hospital, Bristol
  - University Hospital of Llandough, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Dumfries and Galloway Royal Infirmary, Dumfries
  - Western General, Edinburgh
  - Northwick Park Hospital, Harrow
  - St James's University Hospital, Leeds
  - Royal Liverpool Hospital, Liverpool
  - Royal Marsden Hospital, London
  - Borders General Hospital, Melrose
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Peterborough City Hospital, Peterborough
  - Poole Hospital, Poole
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Singleton Hospital, Swansea
  - Arrowe Park Hospital, Upton
  - Thomas Linacre Centre, Wigan

IPD SHARING:
Plan to Share IPD: Undecided